CLINICAL TRIAL: NCT05143983
Title: Perception of Music and Facial and Vocal Emotions in a Population With and Without Depression
Acronym: MusInDep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-A01916-35
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2021-11

CONDITIONS: Depression
Keywords: music; depression; elderly; Emotion perception
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Two groups of participants will be recruited: depressed patients and healthy controls. Each of these groups will be divided in two arms: one group listening to positive music at the first testing visit and neutral music at the second one, and the other group being exposed to positive and neutral conditions in the reverse order.
Who Masked: Participant
Masking Description: Subjects masked from the study hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- depressed subjects, positive valence music listening at first (Active Comparator): patients with major depressive disorder will be recruited and will complete 3 cognitive tasks after listening to positive musical excepts (3 minutes)
  Interventions: Behavioral: Positive valence music
- depressed subjects, neutral valence music listening (Other): patients with major depressive disorder will be recruited and will complete 3 cognitive tasks after listening to neutral valence musical excepts (3 minutes)
  Interventions: Behavioral: Neutral valence music
- healthy controls, positive valence music listening (Other): healthy individuals will be recruited and will complete 3 cognitive task after listening to positive valence musical excepts (3 minutes)
  Interventions: Behavioral: Positive valence music
- healthy controls, neutral valence music listening (Other): healthy individuals will be recruited and will complete 3 cognitive task after listening to neutral valence musical excepts (3 minutes)
  Interventions: Behavioral: Neutral valence music

INTERVENTIONS:
Behavioral: Positive valence music — Subjects will have to listen to 3 minutes of unfamiliar musical excerpts, with positive valence characteristics (fast tempo, major key). They will be told to listen carefully in order to then answer a short questionnaire. The listening will be followed by an liking scale (from 1 : not liked at all, to 5 : liked a lot) and a familiarity scale (from 1 : not familiar at all, to 5 : very familiar).
  Arms: depressed subjects, positive valence music listening at first; healthy controls, positive valence music listening
Behavioral: Neutral valence music — Subjects will have to listen to 3 minutes of unfamiliar musical excepts with neutral valence. They will be told to listen carefully in order to then answer to a short questionnaire. The listening will be followed by a liking scale (from 1 : not liked at all, to 5 : liked a lot) and a familiarity scale (from 1 : not familiar at all, to 5 : very familiar).
  Arms: depressed subjects, neutral valence music listening; healthy controls, neutral valence music listening

SUMMARY:
Depressed subjects display a cognitive bias of information processing and emotional self-regulation, which reinforces negative experiences more than positive ones, known as the negativity bias. The link between depressive disorder and negativity bias has been much studied in terms of genetic, neurobiology, structural and functional neuroanatomy and cognitive sciences. It has been admitted that depressed subjects show impairment of facial expressions and prosody recognition, and of implicit memory.

Induction of depressive or elated mood with musical excerpts listening in healthy subjects influences facial emotions perception, respectively by reducing or enhancing recognition skills. However, no study to date already explored the interest of music-induced positive mood for alleviating negativity bias in depressed elderly population.

Main objective : to assess the impact of exposure to positive valence musical excerpts, on evaluation of facial emotions intensity, in a population of elderly patients hospitalized for depression, compared to neutral valence music listening.

Secondary objectives : to assess the impact of exposure to positive valence musical excerpts, on facial and vocal emotions recognition, and on implicit memory of faces, compared to neutral valence music listening.

The same methodology is also applied in a sample of control participants over 65 years to study the mood induction effect by music in elderlies.

DETAILED DESCRIPTION:
The duration of the study, from first to last included subject, is estimated at 6 months, from January to June 2022. Each subject will participate for a period of 5 to 10 days.

Depressed group subjects will be pre-selected from all consecutive patients hospitalized or seen in consultation in geronto-psychiatric ward at Centre Hospitalier Le Vinatier, who agreed to participate in research. Patients will pass a basic cognitive task (MMSE) during the inclusion visit.

Healthy controls will be selected from relatives of patients admitted in Centre Hospitalier Le Vinatier, who agreed to participate in research.

Once included, subjects will be randomized, and will remain blind to study hypotheses until the study end.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women between the ages of 18 and 60 years old
* Major depressive episode of moderate to strong intensity, according to DSM-5 criteria, diagnosed by a Psychiatrist for subjects with depression ; GDS < 5 for healthy subjects
* Being fluent in French

Exclusion Criteria:

* - Neurodegenerative disorder
* Cognitive impairments (MMSE<26)
* Sensory loss not sufficiently corrected, compromising the perception of oral instructions or visual or auditory stimuli
* Impairment of awareness or attentional abilities restricting completion of cognitive tasks lasting 40 minutes.

And for Patients with depressive episode:

* Psychotic or catatonic features of current depressive episode
* Comorbid psychiatric disorder other than major unipolar depressive or anxiety disorders
* Current treatment by electroconvulsive therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Emotional intensity score of facial expressions, rated by participants | up to 9 days
  This intensity score will be calculated for a subject as the mean of intensity scores (from 1 to 5) attributed to negative faces and reverse intensity scores attributed to positive faces. This will give a "negativity score". The higher this score, the more negative emotions are judged as intense and the less positive emotions are judged as intense. This measurement will be collected by a computerized interface in two different sessions, one for each experimental condition.

SECONDARY OUTCOMES:
Emotions recognition | up to 7 days
  Percentage of correct answers to facial and vocal emotion recognition
Implicit memory | 1 day
  Percentage of identification of previously presented faces with positive expression

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel DOREY, MD, PHD, Principal Investigator — CH le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No